CLINICAL TRIAL: NCT02125773
Title: CCTG 599: Pre-exposure Prophylaxis Accessibility Research and Evaluation (PrEPARE) 2
Brief Title: Pre-exposure Prophylaxis Accessibility Research and Evaluation 2
Acronym: PrEPARE2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Sheldon Morris, Clinical Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CCTG 599
Record Dates: First submitted 2014-04-25; First posted 2014-04-29 (Estimated); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: PrEP Uptake; HIV Seronegativity
Keywords: PrEP; Risk score; Self-perception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Informed Risk Score (Experimental): Subjects in the intervention arm will receive an estimate of their risk of HIV infection as estimated by the UCSD calculator.
  Interventions: Behavioral: Informed Risk Score
- Control (No Intervention): Subjects in the control arm will not be provided with the results of the risk calculators.

INTERVENTIONS:
Behavioral: Informed Risk Score — Subjects in the intervention arm will receive an estimate of their risk of HIV infection as estimated by the UCSD calculator. The risk of HIV infection will be based on the subject's responses to the self-reported sexual risk questionnaire and the risk of HIV infection in one year will be extrapolated based on continuation of the same risk behavior. The subjects will also be provided the calculated risk if they were to take PrEP. Subjects in the control arm will not be provided with the results of the risk calculators. Both arms will receive standard of care risk reduction education and information sheets about PrEP.
  Arms: Informed Risk Score

SUMMARY:
This study is a controlled, un-blinded, two-arm, randomized (1:1) clinical trial to determine if providing high-risk subjects with a calculated risk score changes the likelihood of pre-exposure prophylaxis (PrEP) uptake.

DETAILED DESCRIPTION:
All men who have sex with men (MSM) and male-to-female transgender individuals who have sex with men who present to TNC for HIV testing and are at risk for HIV will be offered enrollment in this study (see study schema). Upon enrollment, subjects will be given an Ipad-based computerized questionnaire that assesses their risk perception, demographics, risk behavior, and perception of whether they are a candidate for PrEP. Upon completion of the survey they will be randomized into 1 of 2 arms. Subjects in the intervention arm will receive the results of their risk score based on a risk calculator developed at UCSD and the Center for Disease Control and Prevention's tool for Assessing Risk for Contracting HIV (ARCH, formerly known as the HIV Incidence Risk Index for MSM, or HIRI-MSM), whereas subjects in the control arm will not receive this information. Both groups will receive standard risk reduction counseling. Subjects will be contacted by phone 2 months after enrollment to determine whether they initiated PrEP or not, to re-assess their risk perception, and to provide a link to a final online survey. If subjects have not completed the survey 4 weeks after being provided with the link, they will receive a text-message reminder.

The analysis of the data will begin 12 weeks after the last study subject is enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Man or transgender M to F who has sex with men.
* Age 18 years or older.
* Subjects must have substantial ongoing risk of acquisition of HIV as evident by one or more of the following: One or more episode of unprotected anal intercourse with a HIV-infected partner or a partner with unknown HIV status within the last 6 months
* Negative for HIV infection by rapid HIV test

Exclusion Criteria:

* Unable to give informed consent.
* Signs or symptoms suggestive of acute HIV infection
* Any other reason or condition that in the opinion of the investigator would interfere with participation, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-02-19 (Actual); Primary Completion 2017-10-09 (Actual); Study Completion 2019-11-08 (Actual)

PRIMARY OUTCOMES:
PrEP uptake between informed vs not-informed of risk score | 12 Weeks
  To compare the proportion of subjects that initiate PrEP between subjects who were informed of their calculated HIV risk score to that of subjects who were not informed of their calculated risk score

CONTACTS AND LOCATIONS:
Overall Officials: Jill Blumenthal, MD, Principal Investigator — CCTG, UCSD AVRC
Locations (1):
- University of California, San Diego, San Diego, California, United States